CLINICAL TRIAL: NCT06428890
Title: Effect of 7 Days of Grape Seed Extract Supplementation on Cold Pressor Test and Muscle Metaboreflex in Individuals With Elevated and Stage 1 Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Baptist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 030-2223-EXP
Record Dates: First submitted 2024-05-15; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Prehypertension
MeSH Terms: conditions — Prehypertension | interventions — Grape Seed Extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Supplementation with Grape Seed Extract (Experimental): Participants received the supplement (600 mg, capsules) via cross-over design for 7 days
  Interventions: Dietary Supplement: Grape Seed Extract; Dietary Supplement: Placebo
- Placebo (Placebo Comparator): Participants received the placebo (600 mg, capsules) via cross-over design for 7 days
  Interventions: Dietary Supplement: Grape Seed Extract; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Grape Seed Extract — dietary supplements that rich in polyphenolic compounds
Dietary Supplement: Placebo — Starch

SUMMARY:
This study aimed to assess the effect of the supplementation with grape seed extract (GSE) on blood pressure during static handgrip exercise and muscle metaboreflex in individuals with elevated and state 1 hypertension.

DETAILED DESCRIPTION:
Muscle metatoreflex (MMR) has been known to play an important role in adjusting hemodynamic responses during exercise. The reflex increases sympathetic activity to heart and blood vessels to increase blood supply to contracting skeletal muscles. On the other hand, studies demonstrated that abnormal cardiovascular responses occurred by the overactive MMR in pathological conditions such as hypertension, diabetes, and congestive heart failure. Excessive blood pressure (BP) responses to exercise induce cardiovascular events such as stroke, heart attack, and coronary artery disease. Previously, a study found that dietary supplementation with grape seed extract (GSE) reduced BP response to dynamic exercise in individuals with elevated and stage 1 hypertension (ES1H) and associated with peripheral vasodilation. However, mechanisms underlying this phenomenon are not clear. Purpose: therefore, the purpose of this study is to investigate whether chronic dietary supplementation with GSE can decrease BP responses to exercise and this observation is associated with reduced MMR. Methods: 12 ES1H males were studied. Changes in cardiac output (Q), mean arterial pressure (MAP) and total peripheral resistance (TPR) were compared between the GSE and placebo supplementations during static handgrip exercise (SHE) and post exercise muscular ischemia (PEMI). Participants completed 3 min of SHE at 40% of MVC followed by 2 min of PEMI.

ELIGIBILITY:
Inclusion Criteria:

* systolic blood pressure: 120-139 mmHg and/or a diastolic blood pressure: 80-89 mmHg

Exclusion Criteria:

* taking medications that could affect cardiovascular function or BP

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
heart rate (bpm) | 5 minutes, 3 minutes, and 2 minutes, respectively.
  measured these variables at rest and during static handgrip exercise and muscle metaboreflex
stroke volume (ml) | 5 minutes, 3 minutes, and 2 minutes, respectively.
  measured these variables at rest and during static handgrip exercise and muscle metaboreflex
cardiac output (l/min) | 5 minutes, 3 minutes, and 2 minutes, respectively.
  measured these variables at rest and during static handgrip exercise and muscle metaboreflex
systolic blood pressure (mmHg) | 5 minutes, 3 minutes, and 2 minutes, respectively.
  measured these variables at rest and during static handgrip exercise and muscle metaboreflex
diastolic blood pressure (mmHg) | 5 minutes, 3 minutes, and 2 minutes, respectively.
  measured these variables at rest and during static handgrip exercise and muscle metaboreflex
total peripheral resistance (mmHg/l/min) | 5 minutes, 3 minutes, and 2 minutes, respectively.
  measured these variables at rest and during static handgrip exercise and muscle metaboreflex

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Kyung Kim, Ph.D., Principal Investigator — California Baptist University
Locations (1):
- California Baptist University, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: No
This study needs the Institutional Research Board (IRB) and participant's approvals to share the data. Without the approval, the data collected from this study will not be shared.